CLINICAL TRIAL: NCT00767676
Title: Evaluation of the Contact Sensitization Potential of 828 Ointment in Normal Healthy Adults
Brief Title: Contact Sensitization Potential of 828 Ointment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: 828-101-09-011
Record Dates: First submitted 2008-10-04; First posted 2008-10-07 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteers
Keywords: Contact sensitization; Healthy Adult Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Device: HP828-101

INTERVENTIONS:
Device: HP828-101 — Nine topical patch applications over 3 weeks, rest period of 2 weeks and challenge after 48 hours.

SUMMARY:
Contact sensitization by patch applications.

DETAILED DESCRIPTION:
Single site study that will evaluate the contact sensitization potential of 828 ointment by repetitive patch applications to the skin of normal, healthy volunteers.

ELIGIBILITY:
1. SUBJECTS 1.1 SUBJECT POPULATION

Subjects will be normal, healthy volunteers of both genders aged 18 to 65 years.

Inclusion Criteria:

Subjects must satisfy all of the following criteria:

1. Subjects must be ambulatory, 18 to 65 years of age and in reasonably good health (no physical required).
2. Subjects may be of any race or skin type provided their skin pigmentation does not interfere with evaluations.
3. Female subjects must be surgically sterile, post-menopausal or using an acceptable method of birth control.
4. Minor deviations in normal medical history not considered to be clinically significant by the investigator and the sponsor will be permitted.
5. Subjects must refrain from sunbathing, using tanning salons, swimming, or using hot tubs during the entire study.
6. Bathing is permitted but subjects must agree to try and keep the patches as dry as possible.
7. Subjects must read and sign the informed consent statement.
8. All females of child bearing potential must agree to take an entry and exit urine pregnancy test

Exclusion Criteria:

Subjects with any of the following conditions are not eligible for participation:

1. Any systemic disease or disorder, complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study (i.e., hepatitis, acute or chronic renal insufficiency).
2. Use of a prescribed pain medication, prescribed or over-the-counter anti-inflammatory drugs, immunosuppressive drugs or prescribed antihistamine medication (steroid nose drops and/or eye drops are permitted). Use of any over-the-counter pain medication that is ingested in quantities exceeding label instructions.
3. Subjects who have received an investigational drug or have participated in a Draize type patch test within the past 28 days or who are currently participating in or plan to enter a clinical trial.
4. A history of non-compliance or subjects who are considered potentially unreliable.
5. A history of skin allergies, including known sensitivity or strong reactions to any cosmetics and/or personal care products, topically prepared medical dressings, tapes, or adhesives.
6. A history of clinically significant skin diseases which may contraindicate participation, including psoriasis, active eczema (at the test sites), atopic dermatitis, and active cancer, even if currently controlled through medication.
7. Current use of topical or oral antibiotics.
8. Use of topical medications at the test area 2 weeks prior to enrollment or any body lotions/oils/creams at the test area for 48 hours prior to enrollment and throughout the trial.
9. Female subjects who are pregnant, stop contraceptive measures, expect to become pregnant or who are breast-feeding.
10. Subjects with any condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
11. Subjects with hematological disorders or immunologic disorders (HIV positive, AIDS, and Systemic Lupus Erythematosus).
12. Subjects with any significant organ abnormality or disorders including gastric ulcer/insulin dependent diabetes.
13. Subjects with any clinically significant illness (sought medical attention, fever, took prescription medication) within the 4 weeks prior to study entry.
14. History of asthma, chronic bronchitis or any other bronchospastic condition that requires medication.
15. Anticipated change in the use of a systemic medication during the study that may affect the conduct or outcome of the study. Subjects must be stabilized on these medications for a least one month prior to receiving study drug and continue same regimen throughout the study.
16. Bilateral mastectomy for cancer involving removal of lymph nodes.
17. Treatment of any type of cancer within the last six months.
18. The Investigator may declare any subject ineligible for a sound medical reason.
19. Subjects with allergies/known sensitivities to any of the ingredients of the test article.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint; Innes Cargill, PhD, Study Director — Healthpoint
Locations (1):
- RCTS, Inc., Irving, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult volunteers, 18 years of age and older
Groups:
- HP828-101: HP828-101 : Nine topical patch applications, each the approximate size of a nickel, over 3 weeks, rest period of 2 weeks and challenge after 48 hours.
Period: Overall Study
Arm/Group | HP828-101
Started | 259
Completed | 205
Not Completed | 54
Not completed — Investigator error | 54

BASELINE CHARACTERISTICS:
Groups:
- HP828-101: HP828-101 : Nine topical patch applications over 3 weeks, rest period of 2 weeks and challenge after 48 hours.
Arm/Group | HP828-101
Number analyzed (Participants) | 259
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 256
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177
  Male | 82
Region of Enrollment [Number; unit: participants]
  United States | 259

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Exhibited a Score Less Than 1.5 on the Jordan-King Scale
Description: To qualify for the claim of a reduced sensitization potential, all subjects completing the study could exhibit a value of no more than 1.5 on the Jordan-King Scale [scale is 0 (no visible reaction) to 5 (severe erythema)]
  No statistical analyses were performed.
Time Frame: 7 weeks
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | HP828-101
Number analyzed (Participants) | 205
participants | 205

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | HP828-101
Serious Adverse Events (participants affected / at risk) | 0/259
Other Adverse Events (participants affected / at risk) | 0/259

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less